CLINICAL TRIAL: NCT05355558
Title: A Novel Functional Imaging Technique With FLT-PET/MRI For Staging, Response Assessment and Radiation Treatment Planning in Cervix Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LEGEND19
Record Dates: First submitted 2022-01-12; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2021-09

CONDITIONS: Image, Body; Cervix Cancer
Keywords: PET/MRI; Imaging technique; Cervix Cancer; FLT PET radiotracer; Response assessment; Radiation treatment
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]FLT-PET/MRI body scan (Experimental)
  Interventions: Diagnostic Test: [18F]FLT-PET/MRI body scan

INTERVENTIONS:
Diagnostic Test: [18F]FLT-PET/MRI body scan — [18F]FLT-PET/MRI body scan will be done at
  * Visit 2 (Baseline-Pre-Treatment FLT-PET/MRI) which will occur between 1 to 28 days prior to initiation of radiotherapy.
  * Visit 3 (During Treatment FLT-PET/MRI) which will occur between week 4 to week 5 of External Beam Radiotherapy (before brachytherapy).
  At these visits:
  * Obtain vital signs and weight in kg before FLT administration.
  * Record the dose of FLT received and injected. (**specify dose: 1mCi per 10kg. Maximum injected dose: < 10mCi per patient.)
  * Place one (1) IV catheters into the participant's arm vein to inject the bolus of FLT.
  * Perform a saline flush following the FLT injection.
  * Body PET/MRI will be performed after FLT injection.
  * Time of injection of FLT and time of scan will need to be recorded.

SUMMARY:
This pilot study aims to monitor early tumour response based on [18F]FLT-PET/MRI scans and to determine the feasibility of personalised radiotherapy to spare active bone marrow areas identified by [18F]FLT-PET/MRI. Bone marrow within the pelvis will be outlined by employing 18FLT PET to identify active BM within bony structures. Subsequently, treatment plans with various conformal radiotherapy techniques will be generated with different optimization approaches toward bone marrow while ensuring adequate tumor coverage.

Dosimetric comparison amongst plans will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent, with the understanding that consent may be withdrawn at any time without prejudice
* Histologically or cytologically confirmed cervical carcinoma
* FIGO staged IB to IVA
* Underwent MRI pelvis
* Underwent FDG-PET/CT or MRI abdomen or CT thorax and abdomen or Chest X ray for routine staging
* Planned for radical radiotherapy with or without chemotherapy
* No distant metastasis in staging work up
* ECOG 0-2
* Age 21 or over (no upper age limit)

Exclusion Criteria:

* Patients scheduled for neoadjuvant chemotherapy
* Patients with previous hysterectomy or radiotherapy to the pelvis
* Patients who are pregnant or lactating
* Patients who do not meet the above mentioned inclusion criteria
* Patients who refuse to give and/or sign the informed consent
* Patients who currently have a pacemaker
* Patients who have a history of serious adverse events related to a previous MRI or PET/CT
* Patients who are unable to undergo MRI scanning
* Patients with a known allergy against any component of the contrast enhancing agent
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow up schedule; these conditions should be discussed with the patient before registration in the trial.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of [18F]FLT-PET/MRI imaging for early prediction of treatment by comparison of changes in baseline SUV uptake at Week 4-5 of External Beam Radiotherapy | Baseline (1 to 28 days before prior initiation of radiotherapy) and Week 4 - 5 of External Beam Radiotherapy (before brachytherapy)

SECONDARY OUTCOMES:
Compare SUV uptake of FLT with FDG PET at diagnosis | Baseline, 1 to 28 days before prior initiation of radiotherapy and Week 4 - 5 of External Beam Radiotherapy (before brachytherapy)
Compare SUV uptake of FLT before and after chemoRT | Baseline, 1 to 28 days before prior initiation of radiotherapy and Week 4 - 5 of External Beam Radiotherapy (before brachytherapy)
To compare differences in tumor and regional staging between PET/MRI, PET/CT and MRI scans, determined from the tumor size and extent of local involvement | Baseline (1 to 28 days before prior initiation of radiotherapy) and Week 4 - 5 of External Beam Radiotherapy (before brachytherapy)
Assess the feasibility of PET/MRI in the radiation treatment planning workflow with respect to the adequacy of image quality and image fusion of PET/MRI data with the treatment planning CT for marrow sparing RT plan | Through patient treatment completion, an average of 3 months
Compare changes in stimulated radiation treatment volume when derived from PET/MRI vs PET/CT vs MRI | Baseline, 1 to 28 days before prior initiation of radiotherapy and Week 4 - 5 of External Beam Radiotherapy (before brachytherapy)
Compare VMAT versus IMRT versus proton versus tomotherapy for best marrow sparing plan | Baseline, 1 to 28 days before prior initiation of radiotherapy and Week 4 - 5 of External Beam Radiotherapy (before brachytherapy)
To determine the correlation of [18F]FLT parameters as baseline, during treatment and change in [18F] FLT parameters with clinical outcome and response | Baseline, 1 to 28 days before prior initiation of radiotherapy and Week 4 - 5 of External Beam Radiotherapy (before brachytherapy)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No